CLINICAL TRIAL: NCT02924571
Title: Prospective, Blinded, Non-randomized Study of Thoracolumbar Spinal Fusion Graft Efficacy: Bone Marrow Aspirate Concentrate and Allograft Versus Recombinant Bone Morphogenetic Protein-2 (BMP)
Brief Title: BMAC & Allograft vs BMP-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-01160
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Spinal Fusion
MeSH Terms: interventions — Transplantation, Homologous; Transplantation, Autologous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Bone Marrow Aspirate Concentrate (BMAC) + Allograft (Experimental): A total of 60, 120, or 180 mL of BMA to be aspirated. BMA is then placed into the Harvest SmartPrep® Bone Marrow Concentrate (BMAC) system and concentrated to a final volume of 10, 20, or 30 mL. The BMAC will then be combined with packed allograft cancellous bone chips using the Harvest Graft Delivery Pack. The allograft bone will be obtained routinely from the bone bank in the operating suite.
  If using Harvest Graft Delivery Kit, the BMAC dosing estimate is as follows (BMAC to graft ratio will be 1:1):
  * 1-level fusion: 10 cc of BMAC from 60 cc of BMA (roughly 10 cc of graft)
  * 2-level fusion: 20 cc of BMAC from 120 cc of BMA
  * 3-level fusion: 20 cc of BMAC from 120 cc of BMA
  * 4-level fusion: 180 cc kit
  * 5-level fusion: 240 cc kit
  If not using Harvest Graft Delivery Kit:
  * Volume of BMAC will be slightly increased (some BMAC will not get directly into hydrating the graft as the BMAC would get lost in the hydration process and left in mixing bowls).
  Interventions: Device: Bone Marrow Aspirate Concentrate (BMAC) + Allograft
- Recombinant Human Bone Morphogenetic Protein-2 (BMP) (Active Comparator): 12 mL BMP will be applied at the surgical site of the interbody fusion using a collagen sponge following manufacturer's directions.
  The BMP kit use per level is as follows:
  * 1 Level Fusion: Extra small kit (1.4 cc)
  * 2 Level Fusion: Small Kit (2.8cc)
  * 3 Level Fusion: (4.2 cc)
  * 4 Level Fusion: Medium Kit (5.6cc)
  * 5 Level Fusion: (7.0 cc)
  Interventions: Device: Recombinant Human Bone Morphogenetic Protein-2 (BMP)
- Autograft (Active Comparator): As per standard of care, the control group will receive 15cc - 45 cc of allograft with autograft and bone marrow aspirate at each level. The iliac crest is the common donor site for autograft. Using the standard technique for anterior lateral fusion, the bone graft will be laid onto the desired site of fusion.
  Interventions: Procedure: Autograft

INTERVENTIONS:
Device: Bone Marrow Aspirate Concentrate (BMAC) + Allograft — Allograft infused with adult stem cells from the bone marrow aspirate harvested from the iliac crest. Harvest BMAC System delivers high stem cell concentration to the graft site.
  Other Names: Harvest BMAC System
  Arms: Bone Marrow Aspirate Concentrate (BMAC) + Allograft
Device: Recombinant Human Bone Morphogenetic Protein-2 (BMP) — INFUSE rhBMP-2 Bone Graft used according to its approved FDA labels, both from an anterior approach using titanium cages as well as from a posterior interbody approach using polyetheretherketone (PEEK) cages.
  Other Names: INFUSE rhBMP-2
  Arms: Recombinant Human Bone Morphogenetic Protein-2 (BMP)
Procedure: Autograft — Autograft with bone marrow aspirate.
  Arms: Autograft

SUMMARY:
The aim of this investigation is to compare the use of bone marrow aspirate concentrate (BMAC) and allograft versus recombinant human bone morphogenetic protein-2 (BMP) versus the gold standard fusion in subjects undergoing elective lumbar spinal fusion with interbody support. The safety and efficacy of the surgical interventions will be evaluated by assessing fusion status and subjects' quality of life outcomes.

DETAILED DESCRIPTION:
This study will be a prospective, randomized clinical study at a single-center, NYU Langone Medical Center. It is intended to compare and evaluate the efficacy of subjects who are either treated with (1) bone marrow aspirate concentrate (BMAC) and allograft or (2) recombinant human bone morphogenetic protein-2 (BMP) or (3) autograft (control) during lumbar spinal fusion with interbody support. The clinical, radiographic, and Health Related Quality of Life (HRQOL) outcomes will be assessed in operatively treated adult spinal degenerative disease patients undergoing lumbar spinal fusion.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years old or older
* Scheduled for elective posterior or anterior and posterior spinal fusion of the thoracolumbar spine with or without anterior interbody support
* Failed at least 6 weeks of conservative care
* No contraindication to BMAC (as per manufacturer)
* Signed consent form

Exclusion criteria:

* Prior lumbar fusion surgery at operative level (prior discectomy and/or laminectomy allowed)
* Incompetent or missing anterior arch at the affected level (e.g. laminectomy, pars defect)
* Currently requires laminectomy at level of surgery
* Facet joints at implant level are absent or fractured
* Post-traumatic vertebral body compromise or acute fracture at implant level
* Body mass Index (BMI) > 40
* Known allergy to titanium
* Paget's disease, osteomalacia, or any other metabolic bone disease
* Use of medications or any drug known to potentially interfere with bone/soft tissue healing (e.g. chronic systemic steroids)
* Unlikely to comply with the follow-up evaluation schedule
* Active malignancy defined as history of invasive malignancy, except if the subject has received treatment and displayed no clinical signs and symptoms for at least five years
* Pregnant or planning to become pregnant during the length of study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Passias, Principal Investigator — NYU Langone Medical Center
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bone Marrow Aspirate Concentrate (BMAC) + Allograft: A total of 60, 120, or 180 mL of BMA to be aspirated. BMA is then placed into the Harvest SmartPrep® Bone Marrow Concentrate (BMAC) system and concentrated to a final volume of 10, 20, or 30 mL. The BMAC will then be combined with packed allograft cancellous bone chips using the Harvest Graft Delivery Pack. The allograft bone will be obtained routinely from the bone bank in the operating suite.
  If using Harvest Graft Delivery Kit, the BMAC dosing estimate is as follows (BMAC to graft ratio will be 1:1):
  * 1-level fusion: 10 cc of BMAC from 60 cc of BMA (roughly 10 cc of graft)
  * 2-level fusion: 20 cc of BMAC from 120 cc of BMA
  * 3-level fusion: 20 cc of BMAC from 120 cc of BMA
  * 4-level fusion: 180 cc kit
  * 5-level fusion: 240 cc kit
  If not using Harvest Graft Delivery Kit:
  * Volume of BMAC will be slightly increased (some BMAC will not get directly into hydrating the graft as the BMAC would get lost in the hydration process and left in mixing bowls).
  Bone Marrow Aspirate Concentrate (BMAC) + Allograft: Allograft infused with adult stem cells from the bone marrow aspirate harvested from the iliac crest. Harvest BMAC System delivers high stem cell concentration to the graft site.
- Recombinant Human Bone Morphogenetic Protein-2 (BMP): 12 mL BMP will be applied at the surgical site of the interbody fusion using a collagen sponge following manufacturer's directions.
  The BMP kit use per level is as follows:
  * 1 Level Fusion: Extra small kit (1.4 cc)
  * 2 Level Fusion: Small Kit (2.8cc)
  * 3 Level Fusion: (4.2 cc)
  * 4 Level Fusion: Medium Kit (5.6cc)
  * 5 Level Fusion: (7.0 cc)
  Recombinant Human Bone Morphogenetic Protein-2 (BMP): INFUSE rhBMP-2 Bone Graft used according to its approved FDA labels, both from an anterior approach using titanium cages as well as from a posterior interbody approach using polyetheretherketone (PEEK) cages.
Period: Overall Study
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Started | 20 | 20 | 19
Completed | 19 | 19 | 19
Not Completed | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft | Total
Number analyzed (Participants) | 20 | 20 | 19 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (12.9) | 55.6 (14.2) | 55.9 (13.6) | 56.53 (13.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 10 | 35
  Male | 8 | 7 | 9 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 5 | 14
  Not Hispanic or Latino | 13 | 13 | 10 | 36
  Unknown or Not Reported | 3 | 2 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 7 | 4 | 16
  White | 12 | 10 | 12 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 19 | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Fusion Status at Month 12 Post-Procedure
Description: Fusion status assessed via CT scan by an independent radiologist.
Time Frame: Month 12 Post-Operation
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Participants | 17 | 16 | 16

2. Primary Outcome: Oswestry Disability Index (ODI) Score at Pre-Op Visit
Description: The ODI is a questionnaire used to assess the functional disability caused by low back pain. It consists of 10 questions, each rated on a scale of 0 (none) to 5 (extreme). The scores from the 10 questions are added up to obtain the raw score; the raw score is divided by the maximum possible score (50) and multiplied by 100 to obtain a percentage score, interpreted as follows: 0-20%: Minimal disability, 21-40%: Moderate disability, 41-60%: Severe disability, 61-80%: Crippling disability, and 81-100%: Bedridden or completely disabled.
Time Frame: Pre-Operation Visit (Day 0)
Measure: Mean (Standard Deviation); unit: Percentage score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Percentage score | 64.8 (4.2) | 66.1 (2.5) | 60.2 (2.6)

3. Primary Outcome: ODI Score at Week 6 Follow-Up
Description: as for outcome 2
Time Frame: Week 6 Post-Operation
Measure: Mean (Standard Deviation); unit: Percentage score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Percentage score | 43.5 (3.8) | 40.2 (5.2) | 44.6 (5.1)

4. Primary Outcome: ODI Score at Month 3 Follow-Up
Description: as for outcome 2
Time Frame: Month 3 Post-Operation
Measure: Mean (Standard Deviation); unit: Percentage score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Percentage score | 41.1 (4) | 40.6 (2.5) | 41.8 (2.9)

5. Primary Outcome: ODI Score at Month 6 Follow-Up
Description: as for outcome 2
Time Frame: Month 6 Post-Operation
Measure: Mean (Standard Deviation); unit: Percentage score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Percentage score | 38.2 (3.4) | 40.3 (1.6) | 40.5 (2.1)

6. Primary Outcome: ODI Score at Month 12 Follow-Up
Description: as for outcome 2
Time Frame: Month 12 Post-Operation
Measure: Mean (Standard Deviation); unit: Percentage score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Percentage score | 34.2 (2.2) | 36.5 (2.9) | 36.8 (2.4)

7. Primary Outcome: ODI Score at Month 24 Follow-Up
Description: as for outcome 2
Time Frame: Month 24 Post-Operation
Measure: Mean (Standard Deviation); unit: Percentage score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Percentage score | 28.6 (2.4) | 30.5 (5.1) | 30.9 (3.6)

8. Primary Outcome: Numeric Rating Scale (NRS) - Back Pain Score at Pre-Op Visit
Description: Participants evaluate leg and back pain using a VAS ranging from 0 cm to 10 cm. Lower scores indicate lower levels of pain.
Time Frame: Pre-Operation Visit (Day 0)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 8.1 (0.8) | 7.6 (0.2) | 8.2 (0.3)

9. Primary Outcome: NRS - Back Pain Score at Week 6 Follow-Up
Description: as for outcome 8
Time Frame: Week 6 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 5.3 (1.6) | 5.6 (2.1) | 4.9 (1.9)

10. Primary Outcome: NRS - Back Pain Score at Month 3 Follow-Up
Description: as for outcome 8
Time Frame: Month 3 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 4.8 (1.1) | 5.2 (1.3) | 4.7 (1.6)

11. Primary Outcome: NRS - Back Pain Score at Month 6 Follow-Up
Description: as for outcome 8
Time Frame: Month 6 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 4.7 (1.3) | 5 (1.4) | 4.7 (1)

12. Primary Outcome: NRS - Back Pain Score at Month 12 Follow-Up
Description: as for outcome 8
Time Frame: Month 12 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 4.2 (1.4) | 4.6 (1.7) | 4.4 (1.2)

13. Primary Outcome: NRS - Back Pain Score at Month 24 Follow-Up
Description: as for outcome 8
Time Frame: Month 24 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 4 (1.1) | 4.1 (0.5) | 4.1 (0.9)

14. Primary Outcome: Short Form 12 (SF-12) - Physical Component Summary (PCS) Score at Pre-Op Visit
Description: The SF-12 PCS is a physical component summary score from the Short Form 12 (SF-12) health survey. The PCS portion of the survey comprises 6 items; the item scores are standardized to a final t-score. The final score ranges from 0-100 with a mean of 50. Higher scores indicate greater physical quality of life.
Time Frame: Pre-Operation Visit (Day 0)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 42.5 (0.9) | 47.6 (2.4) | 45.8 (1.8)

15. Primary Outcome: SF-12 - PCS Score at Week 6 Follow-Up
Description: as for outcome 14
Time Frame: Week 6 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 44.5 (1.3) | 48.4 (0.8) | 47.2 (1)

16. Primary Outcome: SF-12 - PCS Score at Month 3 Follow-Up
Description: as for outcome 14
Time Frame: Month 3 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 44.5 (1.3) | 48.4 (0.8) | 47.2 (1)

17. Primary Outcome: SF-12 - PCS Score at Month 6 Follow-Up
Description: as for outcome 14
Time Frame: Month 6 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 49.5 (0.9) | 50.1 (1.2) | 48.8 (1)

18. Primary Outcome: SF-12 - PCS Score at Month 12 Follow-Up
Description: as for outcome 14
Time Frame: Month 12 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 64.2 (1.7) | 61.6 (1.5) | 62.8 (0.9)

19. Primary Outcome: SF-12 - PCS Score at Month 24 Follow-Up
Description: as for outcome 14
Time Frame: Month 24 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 69.4 (0.8) | 67.7 (1.5) | 70.2 (1.2)

20. Primary Outcome: SF-12 - Mental Component Summary (MCS) Score at Pre-Op Visit
Description: The SF-12 MCS is a mental component summary score from the Short Form 12 (SF-12) health survey. The MCS portion of the survey comprises 6 items; the item scores are standardized to a final t-score. The final score ranges from 0-100 with a mean of 50. Higher scores indicate greater mental quality of life.
Time Frame: Pre-Operation Visit (Day 0)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 51.9 (2.6) | 53.4 (1.7) | 55.1 (1.9)

21. Primary Outcome: SF-12 - MCS Score at Week 6 Follow-Up
Description: as for outcome 20
Time Frame: Week 6 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 58.6 (1.1) | 57.5 (0.8) | 58.1 (1.7)

22. Primary Outcome: SF-12 - MCS Score at Month 3 Follow-Up
Description: as for outcome 20
Time Frame: Month 3 Follow-Up Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 58.9 (1.5) | 57.7 (1.3) | 57.8 (1.1)

23. Primary Outcome: SF-12 - MCS Score at Month 6 Follow-Up
Description: as for outcome 20
Time Frame: Month 6 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 63.1 (1.5) | 65.5 (1.2) | 65.2 (0.9)

24. Primary Outcome: Euro-Qol 5-Dimension (EQ-5D) Score at Pre-Op Visit
Description: 5-item self-report questionnaire. Each item describes a different aspect of health: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Participants rank items on a 3-point Likert scale from 1-3: 1 = no problems; 2 = some problems; 3 = extreme problems. The total score is the sum of responses and ranges from 5-15; lower scores indicate better overall health.
Time Frame: Pre-Operation Visit (Day 0)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 10 (1.1) | 11 (1.3) | 10.5 (0.5)

25. Primary Outcome: EQ-5D Score at Week 6 Follow-Up
Description: as for outcome 24
Time Frame: Week 6 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 8.4 (1.3) | 8.1 (0.7) | 9 (1.8)

26. Primary Outcome: EQ-5D Score at Month 3 Follow-Up
Description: as for outcome 24
Time Frame: Month 3 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 8 (2.5) | 7.9 (1.3) | 8.3 (1.7)

27. Primary Outcome: EQ-5D Score at Month 6 Follow-Up
Description: as for outcome 24
Time Frame: Month 6 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 7.6 (1.6) | 7.1 (1.1) | 7.8 (1.3)

28. Primary Outcome: EQ-5D Score at Month 12 Follow-Up
Description: as for outcome 24
Time Frame: Month 12 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 6.9 (1.1) | 7 (1.7) | 7.4 (2)

29. Primary Outcome: EQ-5D Score at Month 24 Follow-Up
Description: as for outcome 24
Time Frame: Month 24 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 7.1 (1) | 7.4 (1.7) | 7 (1.6)

30. Primary Outcome: Pain Catastrophizing Scale (PCS) Score at Pre-Op Visit
Description: Self-report questionnaire containing 13 items that describe different thoughts and feelings that may be associated with pain. Participants rank each item on a Likert scale from 0 (not at all) to 4 (all the time). Scores range from 0 to 52; lower scores indicate lower levels of catastrophic thinking related to pain.
Time Frame: Pre-Operation Visit (Day 0)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 33.6 (2.4) | 35.2 (1.9) | 35.4 (2.8)

31. Primary Outcome: PCS Score at Week 6 Follow-Up
Description: as for outcome 30
Time Frame: Week 6 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 30.4 (1.8) | 29.6 (2.6) | 31.1 (2.4)

32. Primary Outcome: PCS Score at Month 3 Follow-Up
Description: as for outcome 30
Time Frame: Month 3 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 21.5 (2.9) | 25.8 (3.4) | 25.2 (2.5)

33. Primary Outcome: PCS Score at Month 6 Follow-Up
Description: as for outcome 30
Time Frame: Month 6 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 20.6 (3.6) | 22.2 (3.1) | 20.4 (2.6)

34. Primary Outcome: PCS Score at Month 12 Follow-Up
Description: as for outcome 30
Time Frame: Month 12 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 17.3 (2.4) | 19.8 (2.9) | 20.1 (2.1)

35. Primary Outcome: PCS Score at Month 24 Follow-Up
Description: as for outcome 30
Time Frame: Month 24 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 11.3 (2.4) | 14.3 (2.8) | 15.1 (3.1)

36. Primary Outcome: Patient Reported Outcome Measure Information System (PROMIS) Item Bank v1.1 - Pain Interference Score at Pre-Op Visit
Description: 40-item self-report assessing the negative effects of pain on functioning in the range experienced by the vast majority of people who have pain. Participants rank items on a 5-point Likert scale ranging from 0 to 4. The raw score is the sum of responses and ranges from 0-160; lower scores indicate lower interference from pain. The raw score is translated to give a T-score for each participant. The T-score rescales the raw score into a standardized score ranging from 0 to 100, with a mean of 50 and a standard deviation (SD) of 10. Higher T-scores indicate greater interference from pain.
Time Frame: Pre-Operation Visit (Day 0)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 63.2 (3.5) | 65.1 (3.8) | 60.2 (2.8)

37. Primary Outcome: PROMIS Item Bank v1.1 - Pain Interference Score at Week 6 Follow-Up
Description: as for outcome 36
Time Frame: Week 6 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 54.3 (2.7) | 51.1 (2.4) | 55.5 (3.3)

38. Primary Outcome: PROMIS Item Bank v1.1 - Pain Interference Score at Month 3 Follow-Up
Description: as for outcome 36
Time Frame: Month 3 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 50.8 (3.7) | 49.7 (2.5) | 51.4 (2.1)

39. Primary Outcome: PROMIS Item Bank v1.1 - Pain Interference Score at Month 6 Follow-Up
Description: as for outcome 36
Time Frame: Month 6 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 47.4 (2.4) | 47.6 (3.1) | 49.3 (2.8)

40. Primary Outcome: PROMIS Item Bank v1.1 - Pain Interference Score at Month 12 Follow-Up
Description: as for outcome 36
Time Frame: Month 12 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 41.3 (2.8) | 43.7 (2.5) | 43.5 (2.1)

41. Primary Outcome: PROMIS Item Bank v1.1 - Pain Interference Score at Month 24 Follow-Up
Description: as for outcome 36
Time Frame: Month 24 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 33.8 (2.4) | 32.9 (2.9) | 35.4 (2.1)

42. Primary Outcome: PROMIS Scale v1.0 - Pain Intensity 3a Score at Pre-Op Visit
Description: 3-item self-report assessment of how much a participant hurts. Participants rank items on a 5-point Likert scale ranging from 0 (Had no pain) to 4 (Very severe). The raw score is the sum of responses and ranges from 0-12; lower scores indicate lower levels of pain. The raw score is translated to give a T-score for each participant. The T-score rescales the raw score into a standardized score ranging from 0-100, with a mean of 50 and a standard deviation (SD) of 10. Higher T-scores indicate higher intensity of pain.
Time Frame: Pre-Operation Visit (Day 0)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 68.7 (1.8) | 69.5 (1.4) | 70.4 (2.5)

43. Primary Outcome: PROMIS Scale v1.0 - Pain Intensity 3a Score at Week 6 Follow-Up
Description: as for outcome 42
Time Frame: Week 6 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 61.3 (3.4) | 62.4 (2.9) | 60.1 (3.3)

44. Primary Outcome: PROMIS Scale v1.0 - Pain Intensity 3a Score at Month 3 Follow-Up
Description: as for outcome 42
Time Frame: Month 3 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 52.8 (2.7) | 51.9 (2.9) | 54.2 (3.2)

45. Primary Outcome: PROMIS Scale v1.0 - Pain Intensity 3a Score at Month 6 Follow-Up
Description: as for outcome 42
Time Frame: Month 6 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 50.6 (2.5) | 51.3 (1.9) | 52.8 (2.8)

46. Primary Outcome: PROMIS Scale v1.0 - Pain Intensity 3a Score at Month 12 Follow-Up
Description: as for outcome 42
Time Frame: Month 12 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 33.2 (1.9) | 35.5 (1.5) | 38.6 (2.3)

47. Primary Outcome: PROMIS Scale v1.0 - Pain Intensity 3a Score at Month 24 Follow-Up
Description: as for outcome 42
Time Frame: Month 24 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 25.3 (2.4) | 20.1 (2.8) | 23.4 (3.1)

48. Primary Outcome: PROMIS Bank v1.2 - Physical Function Score at Pre-Op Visit
Description: 120-item self-report assessment of physical health, physical function, pain, and fatigue. Participants rank items on a 5-point Likert scale ranging from 0 to 4. The raw score is the sum of responses and ranges from 0-480; lower scores indicate higher levels of physical function. The raw score is translated to give a T-score for each participant. The T-score rescales the raw score into a standardized score ranging from 0 to 100, with a mean of 50 and a standard deviation (SD) of 10. Higher scores indicate greater physical function.
Time Frame: Pre-Operation Visit (Day 0)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 58.9 (2.1) | 60.3 (3.5) | 54.3 (3.1)

49. Primary Outcome: PROMIS Bank v1.2 - Physical Function Score at Week 6 Follow-Up
Description: as for outcome 48
Time Frame: Week 6 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 50.1 (2.5) | 52.6 (1.8) | 51.1 (1.6)

50. Primary Outcome: PROMIS Bank v1.2 - Physical Function Score at Month 3 Follow-Up
Description: as for outcome 48
Time Frame: Month 3 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 48.3 (2.9) | 47.7 (3.2) | 46.5 (2.6)

51. Primary Outcome: PROMIS Bank v1.2 - Physical Function Score at Month 6 Follow-Up
Description: as for outcome 48
Time Frame: Month 6 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 43.6 (2.4) | 44.9 (1.8) | 42.2 (1.7)

52. Primary Outcome: PROMIS Bank v1.2 - Physical Function Score at Month 12 Follow-Up
Description: as for outcome 48
Time Frame: Month 12 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 39.7 (1.9) | 42.4 (1.5) | 40 (1.1)

53. Primary Outcome: PROMIS Bank v1.2 - Physical Function Score at Month 24 Follow-Up
Description: as for outcome 48
Time Frame: Month 24 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 34.1 (2.3) | 37.3 (2.6) | 38 (2)

54. Primary Outcome: PROMIS Bank v2.0 - Mobility Score at Pre-Op Visit
Description: 15-item self-report assessment of activities of physical mobility. Each item is ranked on a 5-point Likert scale ranging from 0 to 4. The raw score is the sum of responses and ranges from 0-60; lower scores indicate higher levels of physical mobility. The raw score is translated to give a T-score for each participant. The T-score rescales the raw score into a standardized score ranging from 0-100, with a mean of 50 and a standard deviation (SD) of 10. Higher T-scores indicate greater physical mobility.
Time Frame: Pre-Operation Visit (Day 0)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 62.1 (2.8) | 60.7 (3.5) | 64.3 (3.2)

55. Primary Outcome: PROMIS Bank v2.0 - Mobility Score at Week 6 Follow-Up
Description: as for outcome 54
Time Frame: Week 6 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 53.6 (3.5) | 55 (2.8) | 56.7 (2.7)

56. Primary Outcome: PROMIS Bank v2.0 - Mobility Score at Month 3 Follow-Up
Description: as for outcome 54
Time Frame: Month 3 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 49.8 (2.6) | 51.1 (2.4) | 53 (2.3)

57. Primary Outcome: PROMIS Bank v2.0 - Mobility Score at Month 6 Follow-Up
Description: as for outcome 54
Time Frame: Month 6 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 47.2 (2.4) | 49.3 (2.8) | 49.8 (2.7)

58. Primary Outcome: PROMIS Bank v2.0 - Mobility Score at Month 12 Follow-Up
Description: as for outcome 54
Time Frame: Month 12 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 42.7 (2.1) | 44 (3.6) | 44.8 (2.5)

59. Primary Outcome: PROMIS Bank v2.0 - Mobility Score at Month 24 Follow-Up
Description: as for outcome 54
Time Frame: Month 24 Post-Operation
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
T-score | 39.5 (2.8) | 41.1 (2.4) | 43 (2.7)

60. Primary Outcome: Length of Operation
Time Frame: Intraoperative Period (Day 0) (typically between 2-7 hours)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
minutes | 324.6 (114.8) | 354.4 (125.3) | 315.7 (133.8)

61. Primary Outcome: Length of Hospital Stay
Time Frame: From admission up to discharge (Up to Year 2 Post-Operation)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Days | 7.1 (4.1) | 8 (4.4) | 7.3 (3.8)

62. Primary Outcome: Blood Loss During Procedure
Time Frame: Intraoperative Period (Day 0) (typically between 2-7 hours)
Measure: Mean (Standard Deviation); unit: Millilitres
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Millilitres | 845.3 (316.7) | 866.1 (286.4) | 833.6 (322.7)

63. Primary Outcome: Number of Participants Using Non-Prescription, Over-the-Counter (OTC) Drugs at Pre-Op Visit
Description: Number of participants taking OTC drugs for pain relief.
Time Frame: Pre-Operation Visit (Day 0)
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Participants | 20 | 20 | 19

64. Primary Outcome: Number of Participants Using Non-Prescription, OTC Drugs at Week 6 Follow-Up
Description: Number of participants taking OTC drugs for pain relief.
Time Frame: Week 6 Post-Operation
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Participants | 20 | 20 | 19

65. Primary Outcome: Number of Participants Using Non-Prescription, OTC Drugs at Month 3 Follow-Up
Description: Number of participants taking OTC drugs for pain relief.
Time Frame: Month 3 Post-Operation
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Participants | 17 | 18 | 18

66. Primary Outcome: Number of Participants Using Non-Prescription, OTC Drugs at Month 6 Follow-Up
Description: Number of participants taking OTC drugs for pain relief.
Time Frame: Month 6 Post-Operation
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Participants | 10 | 12 | 15

67. Primary Outcome: Number of Participants Using Non-Prescription, OTC Drugs at Month 12 Follow-Up
Description: Number of participants taking OTC drugs for pain relief.
Time Frame: Month 12 Post-Operation
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Participants | 9 | 11 | 12

68. Primary Outcome: Number of Participants Using Non-Prescription, OTC Drugs at Month 24 Follow-Up
Description: Number of participants taking OTC drugs for pain relief.
Time Frame: Month 24 Post-Operation
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Participants | 6 | 8 | 8

69. Primary Outcome: Number of Participants With Surgical Complications During Operation
Time Frame: Intraoperative Period (Day 0) (typically between 2-7 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Participants | 0 | 0 | 0

70. Primary Outcome: Number of Participants With Surgical Complications at Week 6 Follow-Up
Time Frame: Week 6 Post-Operation
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Participants | 0 | 0 | 0

71. Primary Outcome: Number of Participants With Surgical Complications at Month 3 Follow-Up
Time Frame: Month 3 Post-Operation
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Participants | 0 | 0 | 0

72. Primary Outcome: Number of Participants With Surgical Complications at Month 6 Follow-Up
Time Frame: Month 6 Post-Operation
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Participants | 0 | 0 | 0

73. Primary Outcome: Number of Participants With Surgical Complications at Month 12 Follow-Up
Time Frame: Month 12 Post-Operation
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Participants | 3 | 4 | 3

74. Primary Outcome: Number of Participants With Surgical Complications at Month 24 Follow-Up
Time Frame: Month 24 Post-Operation
Measure: Count of Participants; unit: Participants
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
Participants | 3 | 4 | 3

75. Primary Outcome: SF-12 - MCS Score at Month 12 Follow-Up
Description: as for outcome 20
Time Frame: Month 12 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 69.4 (0.8) | 67.7 (2.9) | 68.8 (2.5)

76. Primary Outcome: SF-12 - MCS Score at Month 24 Follow-Up
Description: as for outcome 20
Time Frame: Month 12 Post-Operation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
Number analyzed (Participants) | 20 | 20 | 19
score on a scale | 74.2 (2.4) | 75.6 (3.1) | 75.2 (2)

ADVERSE EVENTS:
Time Frame: Month 24 Post-Operation (2 years)
Description: Adverse events related to study will be detected from follow up visits by the patient and during the post-operative period by the principal investigator and co-investigators, through physical exam assessment and reviewing x-rays and CT scans of the subject.
Arm/Group | Bone Marrow Aspirate Concentrate (BMAC) + Allograft | Recombinant Human Bone Morphogenetic Protein-2 (BMP) | Autograft
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 4/20 | 6/20 | 4/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bone Marrow Aspirate Concentrate (BMAC) + Allograft (N=20) | Recombinant Human Bone Morphogenetic Protein-2 (BMP) (N=20) | Autograft (N=19)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Urinary Tract Infection (Renal and urinary disorders) | 1 | 0 | 1
Non-union (Musculoskeletal and connective tissue disorders) | 3 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/71/NCT02924571/Prot_SAP_000.pdf